CLINICAL TRIAL: NCT05012982
Title: Immunometabolic Mechanisms of Blood Flow Restriction Training After Anterior Cruciate Ligament Reconstruction
Brief Title: Immunometabolic Mechanisms of Blood Flow Restriction (BFR) Training After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000030152
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: AirBand

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AirBand followed by uninflated AirBand (Experimental): The order of study days will be randomized. participants will wear an uninflated AirBand as the control intervention during the session in which BFR is not performed,
  Interventions: Device: AirBand; Device: uninflated AirBand
- Uninflated Airbnd followed by AirBand (Experimental): The order of study days will be randomized. participants will wear an uninflated AirBand as the control intervention during the session in which BFR is not performed,
  Interventions: Device: AirBand; Device: uninflated AirBand

INTERVENTIONS:
Device: AirBand — The AirBands will be placed at each of the two training sessions and inflated while an ultrasound probe is placed over the femoral artery. The cuff will be inflated until the artery reaches 60% occlusion. The force will be applied using a wireless Bluetooth signal; participants will not be asked to adjust the device. Participants will be observed by a certified Personal Therapist throughout the training session in order to determine compliance and ensure safety as is standard protocol for a physical therapy session.
Device: uninflated AirBand — Uninflated AirBand will be used as the control intervention during the session in which BFR is not performed

SUMMARY:
This is a crossover phase 4 study to evaluate the impact of blood flow restriction on immunometabolism and gene expression in immune cells in individuals undergoing rehabilitation from anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
This is a single-blind crossover phase 4 study in which participants will be randomized as to the order in which each of two sessions are completed. Although all analyses will be performed by a blinded investigator and participants will wear an uninflated AirBand as the control intervention during the session in which BFR is not performed, participants will likely know which of the two interventions is being performed on which study day.

The AirBands will be placed at each of the two training sessions and inflated while an ultrasound probe is placed over the femoral artery. The cuff will be inflated until the artery reaches 60% occlusion. The force will be applied using a wireless Bluetooth signal; participants will not be asked to adjust the device. Participants will be observed by a certified Personal Therapist throughout the training session in order to determine compliance and ensure safety as is standard protocol for a physical therapy session.

The study team hypothesizes that the BFR will:

* Promote an anabolic immunometabolic signature, reflected in the composition of serum amino acid concentrations and anabolic hormone content
* Enhance anaerobic glycolysis in leukocytes (which has been associated with increased activation in other settings (Marelli-Berg and Jangani, 2018; Pearce and Pearce, 2013))
* Increase leukocyte glucose and pyruvate concentrations, which corresponds to acute energy provision to promote repair

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for two study visits at least 1 week apart
3. All genders, between 18 and 60 years of age
4. In good general health without any underlying medical conditions or prior injury that would place the subject at risk of further injury/illness by participating in the study

Exclusion Criteria:

1. Serious medical conditions including cardiovascular, metabolic (diabetes), rheumatologic, pulmonary, or musculoskeletal.
2. Multiple ligament ruptures or trauma
3. Rheumatoid arthritis or other significant comorbidities
4. Lower extremity vascular pathology, including history of deep vein thrombosis
5. Those with a history of sickle cell trait or disease
6. Use of anticoagulant medications
7. Pregnancy
8. Treatment with another investigational drug or other intervention within one month of Study Day 1
9. Current smoker or tobacco use within 3 months of Study Day 1
10. Febrile illness within 2 weeks of Study Day 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Leukocyte metabolic gene expression | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Gene expression measured by RNAseq. Because of the nature of RNAseq it is not possible to provide a comprehensive list of gene expression that will be measured; however, genes of particular interest include Slc2a3, Slc2a1, Slc2a4, Slc16a3, PC, Pdha1, Acc1, Fasn.
Change in leukocyte substrate preference | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Fractional contributions of glucose and fatty acids to total mitochondrial oxidation will be measured. Each can fuel between 0 and 100% of total mitochondrial oxidation.
Change in amino acids concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Concentrations of all amino acids (alanine, arginine, asparagine, aspartic acid, cysteine, glutamine, glutamate, glycine, histidine, isoleucine, leucine, lysine, methionine, phenylalanine, proline, serine, threonine, tryptophan, tyrosine, valine). Amino acid concentrations may be between 1 and 500 uM. Higher amino acid concentrations may indicate greater muscle breakdown (proteolysis).
Change in glucose concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Glucose may be between 4 and 15 mM. Higher glucose may be indicative of diabetes.
Change in lactate concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Lactate may be between 0.2 and 8 mM. Higher lactate may be indicative of a more intense exercise response.
Change in fatty acid concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Saturated and unsaturated fatty acid concentrations will be measured. Each fatty acid may range from 0 to 5 mM. Increased fatty acid concentrations may be indicative of a greater stress response to exercise.
Change in insulin concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Insulin may range from 0 to 100 uU/ml. Higher insulin may indicate a greater stress response.
Change in glucagon concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Glucagon may range from 0 to 500 pM. Higher glucagon may indicate lower blood glucose concentrations.
Change in catecholamines concentrations | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Epinephrine and norepinephrine (also known as adrenaline and noradrenaline) will be measured. They can range from 0-1000 nM. Higher catecholamide concentrations may indicate a greater stress response to training.

SECONDARY OUTCOMES:
Whether a baseline immunometabolic blueprint predicts the immunometabolic response to resistance training or to BFR. | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Correlation between Outcomes 1-9 at 0, 30 and 60 minutes after training, to Outcomes 1-9 before training
Whether the immunometabolic response correlates with patient-reported soreness following a physical therapy training session. | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  the soreness scale is 0 to 10, with 0 as no pain or soreness and 10 as pain or soreness as bad as it could possibly be.
Change in creatine kinase | Baseline, 0 (immediately at the end of the exercise session), 30, and 60 minutes post exercise
  Creatine kinase concentration

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Perry, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, Milford, Connecticut
  - Gaylord Outpatient Physical Therapy North Haven Clinic, North Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Data will be published, anonymized. Other than publication, the investigators do not plan to share data with other researchers.